CLINICAL TRIAL: NCT05068999
Title: Early Assessment of Shear Wave Elastography Parameters to Assess the Response to Neoadjuvant Chemotherapy in Patients With Invasive Breast Cancer
Brief Title: Shear Wave Elastography Assessment of Neoadjuvant Chemotherapy Response in Patients With Invasive Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Awad Mohamed Ahmed, principle investigator, Assiut University
Other Study IDs: elastography in breast cancer
Record Dates: First submitted 2021-09-25; First posted 2021-10-06 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: shear wave elastography — Shear wave elastography (SWE) is an emerging technology that provides information about the inherent elasticity of tissues by producing an acoustic radiofrequency force impulse, sometimes called an "acoustic wind," which generates transversely-oriented shear waves that propagate through the surrounding tissue and provide biomechanical information about tissue quality. Although SWE has the potential to revolutionize bone and joint imaging, its clinical application has been hindered by technical and artifactual challenges. Many of the stumbling blocks encountered during musculoskeletal SWE imaging are readily recognizable and can be overcome, but progressive advances in technology and a better understanding of image acquisition are required before SWE can reliably be used in musculoskeletal imaging.

SUMMARY:
The aim of this study is to investigate the role of shear wave elastography (SWE) for early assessment of response to neoadjuvant chemotherapy in patients with invasive breast cancer.

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy (NACT) is often used to treat patients with locally advanced breast cancer, large tumor but operable breast cancer, or proven lymph node metastasis. The advantage of NACT is that it can downstage tumor size and increase the rate of breast-conserving surgery as well as providing information on the drug response through assessment of the changes of tumor size . The pathological complete response has consistently been associated with good long-term outcomes, but is achieved in only 10%-20% of cases. Patients who achieve a pathological complete response have a better prognosis than those who do not . Higher rates of pathological complete response can be achieved when selecting for certain breast cancer subtypes and treatment regimens .

Breast cancer is a heterogeneous disease that can be divided into different subtypes by immunohistochemical marker expression or gene expression array data. A new surrogate intrinsic subtype was proposed at the St Gallen meeting to separate luminal A, luminal B (HER2-/HER2+), HER2-enriched, and triple-negative disease . Similarly, tumors may have different prognosis based on their molecular subtypes. The luminal A subtype has a better prognosis than the other subtypes, and the triple-negative subgroup has the worst prognosis . On the other hand, the triple-negative subtype is more sensitive to chemotherapy than luminal A and B breast cancer .

Current techniques available for monitoring response to NACT are positron emission tomography (PET) , sonography, mammography, magnetic resonance imaging (MRI) , and shear wave elastography (SWE) . Conventional sonography and mammography have poor reliability in evaluating the size of residual tumor after chemotherapy . SWE is a recently developed low-cost imaging technique for measuring tissue stiffness in a noninvasive and quantitative manner with high reproducibility . Tissue stiffness has been demonstrated to be significantly correlated with tumor growth as cancer development and progression require extensive reorganization of the extracellular matrix (ECM) . Increased deposition of collagen and other ECM molecules enhances the stiffness of tumoral stroma . Changes in tumor stiffness were significantly greater in patients who had a good response to NACT compared to those resistant to NACT. Breast cancer pre- and post-treatment stiffness obtained from SWE was significantly correlated with the presence of residual cancer . A study in showed that the SWE stiffness measured after 3 cycles of NACT and changes in stiffness from baseline were strongly associated with pCR after 6 cycles. The combination of the post-treatment SWE and grey scale ultrasound has also been shown to be promising for end-of-treatment identification of residual disease and thus response to NACT, with similar accuracies found in assessment by MRI .

Several histopathological classifications are available to categorize the tumor response to NACT. The Miller-Payne grading (MPG) and Residual Disease in Breast and Nodes (RDBN) are systems to assess the pathological response of NACT. MPG provides a five-step scale based on tumor cellularity in the excision/mastectomy specimen compared with the pretreatment core biopsy as follows: grade 1, no reduction in overall cellularity; grade 2, minor (<30%) loss of cellularity; grade 3, estimated 30%-90% reduction in tumor cells; grade 4, >90% loss of tumor cells; and grade 5, no invasive carcinoma (IC); ductal carcinoma in situ may be present.[30] RDBN uses the following formula: level 1, pathological complete response in breast and nodes, without or with carcinoma in situ, and levels 2-4, residual disease in three different amounts, calculated as 0.2 (residual breast tumor size in cm) + the index for the involved nodes (0 for no positive nodes, 1 for 1-4 nodes, 2 for 5-7 nodes, 3 for ≥8 nodes) + the Scarff-Bloom-Richardson grade (1, 2, or 3), which takes into account tumor size, lymph node stage, and histological grade to determine response.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically confirmed infiltrating breast cancer

  * Stage II or stage III disease. Nodal status must be examined by ultrasound, fine needle aspiration, sentinel node biopsy, or FDG-PET scan.
  * Age ≥18
  * Eastern Cooperative Oncology Group performance status ≤1
  * Adequate bone marrow function (ANC >1.5 x 109/l, platelets >100 x 109/l)
  * Adequate hepatic function (ALAT, ASAT and bilirubin <2.5 times upper limit of normal)
  * Adequate renal function (creatinine clearance >50 ml/min)
  * LVEF ≥50% measured by echocardiography or MUGA
  * Absence of any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
  * Absence of any medical condition that would place the patient at unusual risk.
  * Signed written informed consent

Exclusion Criteria:

* • previous radiation therapy or chemotherapy

  * Other malignancy except carcinoma in situ, unless the other malignancy was treated ≥5 years ago with curative intent without the use of chemotherapy or radiation therapy.
  * Current pregnancy or breastfeeding. Women of childbearing potential must use adequate contraceptive protection.
  * Evidence of distant metastases. Evaluation of the presence of distant metastases may include chest X-ray, liver ultrasound, isotope bone-scan, CT-scan of chest and abdomen and/or FDG-PET scan, according to local procedures.
  * Evidence of bilateral infiltrating breast cancer. Evaluation of the presence of bilateral infiltrating breast cancer may include mammography, breast ultrasound and/or MRI breast.
  * Concurrent anti-cancer treatment or another investigational drug.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
shear wave elastography assessment in patients with invasive breast cancer. | from october 2021 to october2022
  measurement of shear wave elastography parameters in patients with invasive breast cancer before and after neoadjuvant chemotherapy and assess the residual cancer burden for each patient.

REFERENCES:
- [Background] Mieog JS, van der Hage JA, van de Velde CJ. Neoadjuvant chemotherapy for operable breast cancer. Br J Surg. 2007 Oct;94(10):1189-200. doi: 10.1002/bjs.5894. PMID 17701939
- [Background] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986
- [Background] von Minckwitz G, Untch M, Blohmer JU, Costa SD, Eidtmann H, Fasching PA, Gerber B, Eiermann W, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Konecny GE, Denkert C, Nekljudova V, Mehta K, Loibl S. Definition and impact of pathologic complete response on prognosis after neoadjuvant chemotherapy in various intrinsic breast cancer subtypes. J Clin Oncol. 2012 May 20;30(15):1796-804. doi: 10.1200/JCO.2011.38.8595. Epub 2012 Apr 16. PMID 22508812
- [Background] Goldhirsch A, Wood WC, Coates AS, Gelber RD, Thurlimann B, Senn HJ; Panel members. Strategies for subtypes--dealing with the diversity of breast cancer: highlights of the St. Gallen International Expert Consensus on the Primary Therapy of Early Breast Cancer 2011. Ann Oncol. 2011 Aug;22(8):1736-47. doi: 10.1093/annonc/mdr304. Epub 2011 Jun 27. PMID 21709140
- [Background] Perou CM, Sorlie T, Eisen MB, van de Rijn M, Jeffrey SS, Rees CA, Pollack JR, Ross DT, Johnsen H, Akslen LA, Fluge O, Pergamenschikov A, Williams C, Zhu SX, Lonning PE, Borresen-Dale AL, Brown PO, Botstein D. Molecular portraits of human breast tumours. Nature. 2000 Aug 17;406(6797):747-52. doi: 10.1038/35021093. PMID 10963602
- [Background] Hu Z, Fan C, Oh DS, Marron JS, He X, Qaqish BF, Livasy C, Carey LA, Reynolds E, Dressler L, Nobel A, Parker J, Ewend MG, Sawyer LR, Wu J, Liu Y, Nanda R, Tretiakova M, Ruiz Orrico A, Dreher D, Palazzo JP, Perreard L, Nelson E, Mone M, Hansen H, Mullins M, Quackenbush JF, Ellis MJ, Olopade OI, Bernard PS, Perou CM. The molecular portraits of breast tumors are conserved across microarray platforms. BMC Genomics. 2006 Apr 27;7:96. doi: 10.1186/1471-2164-7-96. PMID 16643655
- [Background] Carey LA, Dees EC, Sawyer L, Gatti L, Moore DT, Collichio F, Ollila DW, Sartor CI, Graham ML, Perou CM. The triple negative paradox: primary tumor chemosensitivity of breast cancer subtypes. Clin Cancer Res. 2007 Apr 15;13(8):2329-34. doi: 10.1158/1078-0432.CCR-06-1109. PMID 17438091
- [Background] Goldstein NS, Decker D, Severson D, Schell S, Vicini F, Margolis J, Dekhne NS. Molecular classification system identifies invasive breast carcinoma patients who are most likely and those who are least likely to achieve a complete pathologic response after neoadjuvant chemotherapy. Cancer. 2007 Oct 15;110(8):1687-96. doi: 10.1002/cncr.22981. PMID 17722109
- [Background] Straver ME, Glas AM, Hannemann J, Wesseling J, van de Vijver MJ, Rutgers EJ, Vrancken Peeters MJ, van Tinteren H, Van't Veer LJ, Rodenhuis S. The 70-gene signature as a response predictor for neoadjuvant chemotherapy in breast cancer. Breast Cancer Res Treat. 2010 Feb;119(3):551-8. doi: 10.1007/s10549-009-0333-1. Epub 2009 Feb 13. PMID 19214742
- [Background] Kim C, Han SA, Won KY, Hong IK, Kim DY. Early Prediction of Tumor Response to Neoadjuvant Chemotherapy and Clinical Outcome in Breast Cancer Using a Novel FDG-PET Parameter for Cancer Stem Cell Metabolism. J Pers Med. 2020 Sep 17;10(3):132. doi: 10.3390/jpm10030132. PMID 32957507
- [Background] Tudorica A, Oh KY, Chui SY, Roy N, Troxell ML, Naik A, Kemmer KA, Chen Y, Holtorf ML, Afzal A, Springer CS Jr, Li X, Huang W. Early Prediction and Evaluation of Breast Cancer Response to Neoadjuvant Chemotherapy Using Quantitative DCE-MRI. Transl Oncol. 2016 Feb;9(1):8-17. doi: 10.1016/j.tranon.2015.11.016. Epub 2016 Jan 23. PMID 26947876
- [Background] Cho N, Im SA, Park IA, Lee KH, Li M, Han W, Noh DY, Moon WK. Breast cancer: early prediction of response to neoadjuvant chemotherapy using parametric response maps for MR imaging. Radiology. 2014 Aug;272(2):385-96. doi: 10.1148/radiol.14131332. Epub 2014 Apr 13. PMID 24738612
- [Background] Li Q, Xiao Q, Li J, Wang Z, Wang H, Gu Y. Value of Machine Learning with Multiphases CE-MRI Radiomics for Early Prediction of Pathological Complete Response to Neoadjuvant Therapy in HER2-Positive Invasive Breast Cancer. Cancer Manag Res. 2021 Jun 28;13:5053-5062. doi: 10.2147/CMAR.S304547. eCollection 2021. PMID 34234550
- [Background] Evans A, Armstrong S, Whelehan P, Thomson K, Rauchhaus P, Purdie C, Jordan L, Jones L, Thompson A, Vinnicombe S. Can shear-wave elastography predict response to neoadjuvant chemotherapy in women with invasive breast cancer? Br J Cancer. 2013 Nov 26;109(11):2798-802. doi: 10.1038/bjc.2013.660. Epub 2013 Oct 29. PMID 24169359
- [Background] Lee SH, Chang JM, Han W, Moon HG, Koo HR, Gweon HM, Kim WH, Noh DY, Moon WK. Shear-Wave Elastography for the Detection of Residual Breast Cancer After Neoadjuvant Chemotherapy. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S376-84. doi: 10.1245/s10434-015-4828-1. Epub 2015 Aug 22. PMID 26297209
- [Background] Chagpar AB, Middleton LP, Sahin AA, Dempsey P, Buzdar AU, Mirza AN, Ames FC, Babiera GV, Feig BW, Hunt KK, Kuerer HM, Meric-Bernstam F, Ross MI, Singletary SE. Accuracy of physical examination, ultrasonography, and mammography in predicting residual pathologic tumor size in patients treated with neoadjuvant chemotherapy. Ann Surg. 2006 Feb;243(2):257-64. doi: 10.1097/01.sla.0000197714.14318.6f. PMID 16432360
- [Background] Chang JM, Moon WK, Cho N, Yi A, Koo HR, Han W, Noh DY, Moon HG, Kim SJ. Clinical application of shear wave elastography (SWE) in the diagnosis of benign and malignant breast diseases. Breast Cancer Res Treat. 2011 Aug;129(1):89-97. doi: 10.1007/s10549-011-1627-7. Epub 2011 Jun 17. PMID 21681447
- [Background] Bai M, Du L, Gu J, Li F, Jia X. Virtual touch tissue quantification using acoustic radiation force impulse technology: initial clinical experience with solid breast masses. J Ultrasound Med. 2012 Feb;31(2):289-94. doi: 10.7863/jum.2012.31.2.289. PMID 22298873
- [Background] Denis M, Bayat M, Mehrmohammadi M, Gregory A, Song P, Whaley DH, Pruthi S, Chen S, Fatemi M, Alizad A. Update on Breast Cancer Detection Using Comb-Push Ultrasound Shear Elastography. IEEE Trans Ultrason Ferroelectr Freq Control. 2015 Sep;62(9):1644-50. doi: 10.1109/tuffc.2015.007043. PMID 26688871
- [Background] Evans A, Whelehan P, Thomson K, McLean D, Brauer K, Purdie C, Jordan L, Baker L, Thompson A. Quantitative shear wave ultrasound elastography: initial experience in solid breast masses. Breast Cancer Res. 2010;12(6):R104. doi: 10.1186/bcr2787. Epub 2010 Dec 1. PMID 21122101
- [Background] Golatta M, Schweitzer-Martin M, Harcos A, Schott S, Gomez C, Stieber A, Rauch G, Domschke C, Rom J, Schutz F, Sohn C, Heil J. Evaluation of virtual touch tissue imaging quantification, a new shear wave velocity imaging method, for breast lesion assessment by ultrasound. Biomed Res Int. 2014;2014:960262. doi: 10.1155/2014/960262. Epub 2014 Mar 31. PMID 24800257
- [Background] Zhu J, Xiong G, Trinkle C, Xu R. Integrated extracellular matrix signaling in mammary gland development and breast cancer progression. Histol Histopathol. 2014 Sep;29(9):1083-92. doi: 10.14670/HH-29.1083. Epub 2014 Mar 28. PMID 24682974
- [Background] Cox TR, Erler JT. Remodeling and homeostasis of the extracellular matrix: implications for fibrotic diseases and cancer. Dis Model Mech. 2011 Mar;4(2):165-78. doi: 10.1242/dmm.004077. Epub 2011 Feb 14. PMID 21324931
- [Background] Pickup MW, Mouw JK, Weaver VM. The extracellular matrix modulates the hallmarks of cancer. EMBO Rep. 2014 Dec;15(12):1243-53. doi: 10.15252/embr.201439246. Epub 2014 Nov 8. PMID 25381661
- [Background] Gilkes DM, Bajpai S, Wong CC, Chaturvedi P, Hubbi ME, Wirtz D, Semenza GL. Procollagen lysyl hydroxylase 2 is essential for hypoxia-induced breast cancer metastasis. Mol Cancer Res. 2013 May;11(5):456-66. doi: 10.1158/1541-7786.MCR-12-0629. Epub 2013 Feb 1. PMID 23378577
- [Background] Jing H, Cheng W, Li ZY, Ying L, Wang QC, Wu T, Tian JW. Early Evaluation of Relative Changes in Tumor Stiffness by Shear Wave Elastography Predicts the Response to Neoadjuvant Chemotherapy in Patients With Breast Cancer. J Ultrasound Med. 2016 Aug;35(8):1619-27. doi: 10.7863/ultra.15.08052. Epub 2016 Jun 14. PMID 27302898
- [Background] Evans A, Whelehan P, Thompson A, Purdie C, Jordan L, Macaskill J, Waugh S, Fuller-Pace F, Brauer K, Vinnicombe S. Prediction of Pathological Complete Response to Neoadjuvant Chemotherapy for Primary Breast Cancer Comparing Interim Ultrasound, Shear Wave Elastography and MRI. Ultraschall Med. 2018 Aug;39(4):422-431. doi: 10.1055/s-0043-111589. Epub 2017 Sep 21. PMID 28934812
- [Background] Evans A, Whelehan P, Thompson A, Purdie C, Jordan L, Macaskill J, Henderson S, Vinnicombe S. Identification of pathological complete response after neoadjuvant chemotherapy for breast cancer: comparison of greyscale ultrasound, shear wave elastography, and MRI. Clin Radiol. 2018 Oct;73(10):910.e1-910.e6. doi: 10.1016/j.crad.2018.05.030. Epub 2018 Jul 3. PMID 29980324
- [Background] Ogston KN, Miller ID, Payne S, Hutcheon AW, Sarkar TK, Smith I, Schofield A, Heys SD. A new histological grading system to assess response of breast cancers to primary chemotherapy: prognostic significance and survival. Breast. 2003 Oct;12(5):320-7. doi: 10.1016/s0960-9776(03)00106-1. PMID 14659147
- [Background] Chollet P, Amat S, Belembaogo E, Cure H, de Latour M, Dauplat J, Le Bouedec G, Mouret-Reynier MA, Ferriere JP, Penault-Llorca F. Is Nottingham prognostic index useful after induction chemotherapy in operable breast cancer? Br J Cancer. 2003 Oct 6;89(7):1185-91. doi: 10.1038/sj.bjc.6601258. PMID 14520443
- [Background] Chollet P, Abrial C, Durando X, Thivat E, Tacca O, Mouret-Reynier MA, Leheurteur M, Kwiatkowski F, Dauplat J, Penault-Llorca F. A new prognostic classification after primary chemotherapy for breast cancer: residual disease in breast and nodes (RDBN). Cancer J. 2008 Mar-Apr;14(2):128-32. doi: 10.1097/PPO.0b013e31816bdea2. PMID 18391619
- [Background] Abrial SC, Penault-Llorca F, Delva R, Bougnoux P, Leduc B, Mouret-Reynier MA, Mery-Mignard D, Bleuse JP, Dauplat J, Cure H, Chollet P. High prognostic significance of residual disease after neoadjuvant chemotherapy: a retrospective study in 710 patients with operable breast cancer. Breast Cancer Res Treat. 2005 Dec;94(3):255-63. doi: 10.1007/s10549-005-9008-8. PMID 16267618